CLINICAL TRIAL: NCT05069597
Title: A Phase 4 Study to Assess Symptoms of Exocrine Pancreatic Insufficiency in Subjects With Cystic Fibrosis or Chronic Pancreatitis Treated With Creon® (Pancrelipase) With an Alternate Source of Active Pharmaceutical Ingredient
Brief Title: Study to Evaluate Symptoms of Exocrine Pancreatic Insufficiency in Adult Participants With Cystic Fibrosis or Chronic Pancreatitis Treated With Creon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: M21-432
Record Dates: First submitted 2021-09-27; First posted 2021-10-06 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis; Chronic Pancreatitis
Keywords: Cystic Fibrosis; Chronic Pancreatitis; Exocrine Pancreatic Insufficiency; Creon; Pancrelipase
MeSH Terms: conditions — Cystic Fibrosis; Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Run-in Period: Creon-ABT (Experimental): Participants will receive Creon-ABT daily for 28 days.
  Interventions: Drug: CREON
- Treatment Period: Creon-AAPIS (Experimental): Participants will receive Creon-AAPIS daily for 85 days.
  Interventions: Drug: CREON

INTERVENTIONS:
Drug: CREON — Capsule; Oral
  Other Names: Pancrelipase

SUMMARY:
Exocrine pancreatic insufficiency (EPI) is a condition that is caused by the inadequate pancreatic enzymes needed for normal digestion and is commonly associated with a wide range of chronic diseases, including cystic fibrosis (CF), chronic pancreatitis (CP), and pancreatic cancer. This study will assess clinical symptoms when participants with CF or CP are treated with Creon with alternate source of active drug.

Creon is an approved drug for the treatment of EPI. This study is subject-blinded which means participants will not know the source of the study drug they are given. Approximately 30 adult participants with CF or CP will be enrolled at approximately 15 sites across the Unites States.

Participants will receive oral capsules of CREON for 113 days and will be followed for 30 days.

Participants will attend regular visits during the study at a hospital or clinic or via telemedicine. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of cystic fibrosis (CF) or chronic pancreatitis (CP).
* Previous diagnosis of exocrine pancreatic insufficiency (EPI) that is currently clinically controlled.
* Total Symptom Score (TSS) < 1.8 on Pancreatic Exocrine Insufficiency Questionnaire (PEI-Q) at Screening.

Exclusion Criteria:

- Malignancy involving the digestive tract in the last 5 years, or other significant disease or medical condition that may interfere with EPI symptom assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (21):
  - Velocity Clinical Research /ID# 231076, Mobile, Alabama
  - Valley Children's Hospital /ID# 231452, Madera, California
  - University of Florida - Archer /ID# 233411, Gainesville, Florida
  - Atlantic Medical Research /ID# 239568, Margate, Florida
  - University of Miami, Miller School of Medicine /ID# 239415, Miami, Florida
  - GI Pros /ID# 239486, Naples, Florida
  - Central FL Pulmonary Orlando /ID# 245863, Orlando, Florida
  - Asr, Llc /Id# 239566, Nampa, Idaho
  - UMass Chan Medical School /ID# 230476, Worcester, Massachusetts
  - The Curators of the University of Missouri /ID# 233331, Columbia, Missouri
  - Dartmouth-Hitchcock Medical Center /ID# 231633, Lebanon, New Hampshire
  - Albany Medical College-Pulmonary /ID# 250041, Albany, New York
  - NYU Langone Health /ID# 233417, New York, New York
  - Wake Forest Baptist Health /ID# 229537, Winston-Salem, North Carolina
  - University of Cincinnati /ID# 229511, Cincinnati, Ohio
  - UH Cleveland Medical Center /ID# 246065, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 245864, Cleveland, Ohio
  - Options Health Research, LLC /ID# 239535, Tulsa, Oklahoma
  - Baylor College of Medicine Medical Center /ID# 233441, Houston, Texas
  - Univ Texas HSC San Antonio /ID# 239060, San Antonio, Texas
  - West Virginia University Hospitals /ID# 239593, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty participants were enrolled at 13 sites throughout the United States. During the run-in period, 30 participants were treated and completed 28 days of treatment with Creon-ABT.
Pre-assignment Details: One participant failed continuation criteria, with the remaining 29 participants continuing on to the treatment period with Creon-AAPIS. The Per Protocol Population included all enrolled subjects who received at least 1 dose of Creon-AAPIS, had Day 1 (Baseline) PEI-Q scores collected, and had at least one post-baseline PEI-Q scores collected during the Treatment Period (Days 8, 15, 29, and 85).
Groups:
- Run-in: Creon-ABT: Participants received blinded Creon-ABT for the duration of the Run-in Period (28 days) at the same stable individual dose of Creon he/she was on before screening. This assured that the Day 1 assessment reflected the symptoms on stable Creon-ABT use.
- Treatment: Creon-AAPIS: Participants who completed the Run-in Period were assessed for the continuation criteria at Day 1. Blinded Creon-ABT study drug from the Run-In Period was returned, and the participant was dispensed blinded Creon-AAPIS to use at the same stable individual dose per LU of Creon he/she was on before Screening and during the Run-in Period. This assured that the treatment assessments after Day 1 reflect the symptoms on Creon-AAPIS.
Period: Run-in Period (Day -28 to Day 0)
Arm/Group | Run-in: Creon-ABT | Treatment: Creon-AAPIS
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0
Period: Treatment Period (Day 1 to Day 85)
Arm/Group | Run-in: Creon-ABT | Treatment: Creon-AAPIS
Started | 0 | 29
Completed | 0 | 28
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS included all enrolled subjects who received at least 1 dose of study drug of Creon-AAPIS. The FAS was used for the summary of participant disposition, demographics, and baseline characteristics.
Arm/Group | Treatment: Creon-AAPIS
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (16.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Total Symptom Score (TSS) From Day 1 (Baseline) to Days 8, 15, 29, and 85
Description: The Pancreatic Exocrine Insufficiency Questionnaire (PEI-Q) is an 18-item Patient-Reported Outcome (PRO) instrument that assesses EPI symptoms and associated impact over the previous 7 days. All items are scored using a 5-point Likert scale (Not at all to Yes, a lot). The average score for each symptom domain is calculated, ranging from 0 to 4. TSS is calculated from the average of the mean abdominal domain score and the mean bowel movement symptom score. A numerically higher response indicates more severe EPI symptoms. Positive changes from baseline indicate a worsening of symptoms.
Time Frame: Day 1 (baseline), 8, 15, 29, and 85
Population: The Per Protocol Population included all enrolled subjects who received at least 1 dose of study drug of Creon-AAPIS, had Day 1 (Baseline) PEI-Q scores collected, and had at least one post-baseline PEI-Q scores collected during the Treatment Period (Days 8, 15, 29, and 85). The pharmacodynamic endpoints were analyzed in the Per Protocol Population. Number analyzed indicates the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: Creon-AAPIS
Number analyzed (Participants) | 29
score on a scale
  Change from Baseline to Day 8: number analyzed (Participants) | 27
  Change from Baseline to Day 8 | 0.0012 (0.2953)
  Change from Baseline to Day 15: number analyzed (Participants) | 27
  Change from Baseline to Day 15 | 0.0480 (0.4354)
  Change from Baseline to Day 29: number analyzed (Participants) | 27
  Change from Baseline to Day 29 | 0.1506 (0.5396)
  Change from Baseline to Day 85: number analyzed (Participants) | 24
  Change from Baseline to Day 85 | 0.0791 (0.5298)

2. Primary Outcome: Mean Change in Abdominal Symptom Domain Score (ASDS) From Day 1 (Baseline) to Days 8, 15, 29, and 85
Description: The PEI-Q is an 18-item PRO instrument that assesses EPI symptoms and associated impact over the previous 7 days. All items are scored using a 5-point Likert scale (Not at all to Yes, a lot). The average score for each symptom domain is calculated, ranging from 0 to 4. ASDS is the mean abdominal symptom domain score measured by the PEI-Q. A numerically higher response indicates more severe EPI symptoms. Positive changes from baseline indicate a worsening of symptoms.
Time Frame: Day 1 (Baseline), 8, 15, 29, and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: Creon-AAPIS
Number analyzed (Participants) | 29
score on a scale
  Change from baseline to Day 8: number analyzed (Participants) | 27
  Change from baseline to Day 8 | 0.0582 (0.3722)
  Change from baseline to Day 15: number analyzed (Participants) | 27
  Change from baseline to Day 15 | 0.0530 (0.4605)
  Change from baseline to Day 29: number analyzed (Participants) | 27
  Change from baseline to Day 29 | 0.1905 (0.6100)
  Change from baseline to Day 85: number analyzed (Participants) | 24
  Change from baseline to Day 85 | 0.0893 (0.5190)

3. Primary Outcome: Mean Change in Bowel Movement Symptom Score (BMSS) From Day 1 (Baseline) to Days 8, 15, 29, and 85
Description: The PEI-Q is an 18-item PRO instrument that assesses EPI symptoms and associated impact over the previous 7 days. All items are scored using a 5-point Likert scale (Not at all to Yes, a lot). The average score for each symptom domain is calculated, ranging from 0 to 4. BMSS is the mean bowel movement symptom domain score measured by the PEI-Q. A numerically higher response indicates more severe EPI symptoms. Positive changes from baseline indicate a worsening of symptoms.
Time Frame: Day 1 (Baseline), 8, 15, 29, and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: Creon-AAPIS
Number analyzed (Participants) | 29
score on a scale
  Change from Baseline to Day 8: number analyzed (Participants) | 27
  Change from Baseline to Day 8 | -0.0555 (0.3235)
  Change from Baseline to Day 15: number analyzed (Participants) | 27
  Change from Baseline to Day 15 | 0.0432 (0.5240)
  Change from Baseline to Day 29: number analyzed (Participants) | 27
  Change from Baseline to Day 29 | 0.1111 (0.5565)
  Change from Baseline to Day 85: number analyzed (Participants) | 24
  Change from Baseline to Day 85 | 0.0695 (0.7000)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to end of study. The median time participants were followed was 28 days for CREON-ABT and 116 days for CREON-AAPIS.
Arm/Group | Run-in: Creon-ABT | Treatment: Creon-AAPIS
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/29
Other Adverse Events (participants affected / at risk) | 1/30 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in: Creon-ABT (N=30) | Treatment: Creon-AAPIS (N=29)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in: Creon-ABT (N=30) | Treatment: Creon-AAPIS (N=29)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 4 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 6 (9)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 2 (5)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT05069597/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05069597/SAP_001.pdf